CLINICAL TRIAL: NCT00536328
Title: What is the Value of the Use of Validated Questionnaire (Reflux Impact Scale) for Predicting Treatment Success With PPI
Brief Title: What is the Predictive Value of the Reflux Impact Scale
Acronym: PREDICT
Status: Terminated | Type: Observational
Why Stopped: due to very low recruitment. For this reason, there will be no further analysis and reporting of this study.
Sponsor: AstraZeneca (Industry)
Other Study IDs: NL401611
Record Dates: First submitted 2007-09-26; First posted 2007-09-27 (Estimated); Last update posted 2008-07-09 (Estimated); Status verified 2008-07

CONDITIONS: Gastroesophageal Reflux Disease; GERD; Heartburn; Acid Regurgitation; Retrosternal Pain
Keywords: Reflux Impact Scale (RIS); predictive value; treatment success; patient satisfaction; proton pump inhibitor; gastro-esophageal reflux disease; PPU
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn; Patient Satisfaction

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Gastric distress is a common phenomenon in our society. Heartburn and regurgitation occur daily in about 7% of the adult population,weekly 14-20% pf the adults and monthly in 34-44% of adults. The yearly prevalence of recurrent stomach complaints are frequent reason for consulting a primary care physician and are an important reason for using OTC medication. A good diagnosis is important as functional GERD with possible complications such as strictures and Barrett's esophagus or ulcer disease with life threatening complications such as bleeding & perforations. The clinical diagnosis of reflux disease is mainly based on symptom evaluation. This, however, is hindered by the variety of complaints with different etiology. Treatment with a proton pump inhibitor can be used to confirm the diagnosis reflux disease. A major part of the patients with acid related stomach complaints indeed will experience symptom relief after starting PPI therapy. In this view, it is important to identify these patients who will react on treatment with PPI in quick, accurate, non-invasive and cheap manner. The Reflux Impact Scale (RIS) is validated, short, self explanatory questionnaire which asks for the presence & impact of reflux symptoms. The RIS is developed for PCP to aid in the evaluation & selection of these patient who will profit from treatment with PPI. The aim of this present study is to determine which questions of the RIS can be predictive for reaching treatment success with PPI. Treatment success is determined by asking for patients' satisfaction & completion of the McMaster Overall Treatment Evaluation Heartburn questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Patients with symptoms of reflux disease and or regurgitation and/or retrosternal pain probably caused by acid during the previous 7 days and for which treatment with a PPI is started.

Exclusion Criteria:

* Use of PPI and/or H2-receptor antagonist in the month prior to participation in this study.
* Presence of alarm symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting at general practitioner
Sampling Method: Non-Probability Sample
Enrollment: 938 (Estimated)
Dates: Start 2007-10; Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A Sellink, Study Director — AstraZeneca; N van den Berk, Study Chair — AstraZeneca